CLINICAL TRIAL: NCT03449381
Title: A Phase Ia/Ib, Open Label, Multicenter, Dose-escalation Study of BI 907828 (Brigimadlin) in Patients With Advanced or Metastatic Solid Tumors
Brief Title: This Study Aims to Find the Best Dose of BI 907828 (Brigimadlin) in Patients With Different Types of Advanced Cancer (Solid Tumors)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1403-0001; 2017-003210-95 (EudraCT Number)
Record Dates: First submitted 2018-02-12; First posted 2018-02-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — brigimadlin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental)
  Interventions: Drug: BI 907828
- Dose Expansion (Experimental)
  Interventions: Drug: BI 907828

INTERVENTIONS:
Drug: BI 907828 — Film-coated tablet
  Other Names: brigimadlin

SUMMARY:
This study is open to adults with different types of advanced cancer (solid tumors). The purpose of this study is to find out the most suitable dose of BI 907828 (brigimadlin) the participants can tolerate. The most suitable dose is used in the second part to find out whether brigimadlin makes tumors shrink.

In this study, brigimadlin is given to humans for the first time. Brigimadlin is a so-called MDM2 inhibitor that is being developed to treat cancer. Brigimadlin is taken as a tablet. Participants either take a dose of brigimadlin on one day every 3 weeks or on two days every 4 weeks.

The participants are in the study for as long as they benefit from and can tolerate treatment. The doctors regularly check the participants' general health during the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent form ICF in accordance with ICH-GCP and local legislation prior to any trial-specific procedures, sampling, or analyses.
* Pathologically documented, advanced solid tumors.
* Patients fulfilling one or more of the following criteria:

  * Radiologically documented disease progression or relapse
  * Patients who are not eligible to receive standard of care treatments, and for whom no proven treatments exist.
  * Patients with MDM2 amplified sarcomas who require first line treatment (for Ph Ib/dose expansion - Cohort 1 only).
* Patients with MDM2 amplified sarcomas may fulfil any one of the above three criteria to be considered eligible.
* Phase Ia (dose escalation) only:
* Patient has a tumor with either a known TP53 wild type status, or unknown TP53 status, and regardless of MDM2 amplification status, at the time of study entry.
* Phase Ib (expansion phase) only:
* Cohort 1: TP53 wt and MDM2-amplified sarcoma with advanced/metastatic disease at any line of therapy. If TP53 status is not available during screening, the patient may be included with unknown TP53 status if a tissue sample is submitted for central laboratory assessment. If TP53 status cannot be evaluated, the patient may be included if agreed between the Investigator and Sponsor.
* Cohort 2: TP53 wt and MDM2- amplified NSCLC, urothelial, gastric, biliary tract (including cholangiocarcinoma, intra- and extrahepatic biliary tree, gall blander and ampulla of vater) or pancreatic solidPDAC tumors who have had at least one previous line of therapy for advanced/metastatic disease. If TP53 status cannot be evaluated the patient may be included if agreed between the Investigator and Sponsor
* Phase Ia (dose escalation) only:
* Patient with either measurable or non-measurable disease.
* Non-evaluable disease allowed.
* Phase Ib (expansion phase) only:
* At least one target lesion that can be accurately measured per RECIST v.1.1.
* Phase Ia:
* Patient must be willing to undergo blood sampling for PK, pharmacodynamic, biomarker, and PGx analyses.
* Phase Ib:
* Patient must be willing to undergo tumor biopsy sampling for pharmacodynamic analyses and blood sampling for PK, pharmacodynamics, and biomarker analyses.
* Willingness to provide a fresh tumor tissue sample obtained after relapse/ progression during or after prior therapy. In case a fresh biopsy cannot be obtained (e.g. inaccessible lesions or patient safety concern), an archived specimen, collected before screening within 12 months of enrollment, may be submitted. If these requirements cannot be met, then the patient may be allowed to enter the study at Sponsor discretion, after agreement between the Investigator and Sponsor.
* Further inclusion criteria apply

Exclusion Criteria:

* Previous administration of BI 907828 (brigimadlin) or any other MDM2-p53 or MDMX (MDM4)-p53 antagonist.
* Known TP53 mutant tumor.
* Symptomatic metastases from non-brain tumors. Note: Patients with previously treated brain metastases may participate provided they are stable, without evidence of progression by imaging (using the identical imaging modality for each assessment, either MRI or computed tomography (CT) scan), for at least four weeks prior to the first dose of trial treatment, and any neurologic symptoms have returned to baseline; have no evidence of new or enlarging brain metastases. Patients on corticosteroids must have a stable dose for at least 5 days prior to baseline MRI.
* Patients with history of bleeding diathesis.
* Major surgery (major according to the Investigator's assessment) performed within 12 weeks prior to start of study treatment, or planned within 12 months after screening (e.g. hip replacement).
* Any other documented active or suspected malignancy or history of malignancy within 3 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix, or other local tumors considered cured by local treatment.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Phase Ia- Maximum tolerated dose (MTD) based on number of patients with dose limiting toxicities (DLTs) during first treatment cycle | Up to 28 days
Phase Ib - Progression-free survival | Up to 24 months
Phase Ia - Number of patients with DLTs during first treatment cycle (21 days, Arm A; 28 days, Arm B) | Up to 28 days
Phase Ib - Number of patients with DLTs during the first treatment cycle | Up to 28 days

SECONDARY OUTCOMES:
Phase Ia - Cmax: Maximum measured concentration of BI 907828 in plasma | Up to 24 months
Phase Ia - AUC0-∞: Area under the concentration-time curve in plasma over the time interval from 0 extrapolated to infinity | Up to 24 months
Phase Ib - Objective response | Up to 24 months
Phase Ib - Overall survival | Up to 24 months
Phase Ib - Number of patients with Grade ≥3 treatment-related adverse events observed during the entire treatment period | Up to 24 months
Phase Ib - Cmax: Maximum measured concentration of BI 907828 in plasma | Up to 24 months
Phase Ib - AUC0-∞: Area under the concentration-time curve in plasma over the time interval from 0 extrapolated to infinity | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (27):
- United States (9):
  - Sarcoma Oncology Center, Santa Monica, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialists-Sarasota-61670, Sarasota, Florida
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- The Ottawa Hospital, Ottawa, Ontario, Canada
- Rigshospitalet, København, København Ø, Denmark
- Germany (4):
  - Helios Klinikum Berlin-Buch, Berlin
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Universitätsklinikum Tübingen, Tübingen
- Sourasky Medical Center, Tel Aviv, Israel
- National Cancer Center Hospital, Tokyo, Chuo-ku, Japan
- Poland (2):
  - MED POLONIA SP Z O O, Clinical Trials Department,Poznan, Poznan
  - Oncology Center-Maria Sklodowska-Curie Institute, Warsaw
- Severance Hospital, Seoul, South Korea
- Spain (4):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico de Santiago, Santiago de Compostela
- Karolinska Comprehensive Cancer Center, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] LoRusso P, Yamamoto N, Patel MR, Laurie SA, Bauer TM, Geng J, Davenport T, Teufel M, Li J, Lahmar M, Gounder MM. The MDM2-p53 Antagonist Brigimadlin (BI 907828) in Patients with Advanced or Metastatic Solid Tumors: Results of a Phase Ia, First-in-Human, Dose-Escalation Study. Cancer Discov. 2023 Aug 4;13(8):1802-1813. doi: 10.1158/2159-8290.CD-23-0153. PMID 37269344
- See also: Related Info — https://www.mystudywindow.com